CLINICAL TRIAL: NCT04589975
Title: CONVERSION TO OPEN SURGERY IN LAPAROSCOPIC COLORECTAL CANCER RESECTION: PREDICTIVE FACTORS AND ITS IMPACT ON LONG-TERM OUTCOMES. A RETROSPECTIVE COHORT STUDY
Brief Title: Predictive Factors of Conversion in Laparoscopic Colorectal Cancer Resection
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: PFLC
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Surgery; Colorectal Neoplasm; Laparoscopy
Keywords: Laparoscopic surgery, colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscopic surgery

SUMMARY:
Background Laparoscopic resection is the treatment of choice for colorectal cancer. Rates of conversion to open surgery range between 7% and 30% and controversy exists as to the effect of this on oncologic outcomes. The objective of this study was to analyze what factors are predictive of conversion and what effect they have on oncologic outcomes.

Material & Methods From a prospective database of patients undergoing laparoscopic surgery between 2000 and 2018 a uni- and multivariate analyses were made of demographic, pathological and surgical variables together with complementary treatments comparing purely laparoscopic resection with conversions to open surgery. Overall and disease-free survival were compared using the Kaplan-Meier method.

DETAILED DESCRIPTION:
Laparoscopic resection of colorectal cancer is the surgical option of choice provided that established oncologic principles are guaranteed [1-4].

Apart from the well-known advantages of minimally invasive surgery (shorter hospital stays, lower pain levels, faster return of bowel functions and rapid return to normal daily activities) reductions in operative morbidity and mortality have been reported together with oncologic outcomes which are similar to those of open surgery [5-7].

However, reported conversion rates to open surgery are highly variable (7% - 30%) as is the impact of conversion on oncologic outcomes [8-10]). The objectives of this study were to identify the risk factors associated with conversion and to assess their impact on operative morbidity and mortality and long-term oncologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All laparoscopic colorectal neoplasia, laparoscopic resected

Exclusion Criteria:

* Palliative and emergency procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Colorectal cancer patient, surgical resected by laparoscopy
Sampling Method: Probability Sample
Enrollment: 829 (Actual)
Dates: Start 2000-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Conversion to open rate: predictive factors oncological outcomes | 2000-2018

REFERENCES:
- [Background] Colon Cancer Laparoscopic or Open Resection Study Group; Buunen M, Veldkamp R, Hop WC, Kuhry E, Jeekel J, Haglind E, Pahlman L, Cuesta MA, Msika S, Morino M, Lacy A, Bonjer HJ. Survival after laparoscopic surgery versus open surgery for colon cancer: long-term outcome of a randomised clinical trial. Lancet Oncol. 2009 Jan;10(1):44-52. doi: 10.1016/S1470-2045(08)70310-3. Epub 2008 Dec 13. PMID 19071061
- [Background] Fleshman J, Sargent DJ, Green E, Anvari M, Stryker SJ, Beart RW Jr, Hellinger M, Flanagan R Jr, Peters W, Nelson H; Clinical Outcomes of Surgical Therapy Study Group. Laparoscopic colectomy for cancer is not inferior to open surgery based on 5-year data from the COST Study Group trial. Ann Surg. 2007 Oct;246(4):655-62; discussion 662-4. doi: 10.1097/SLA.0b013e318155a762. PMID 17893502
- [Background] Allaix ME, Furnee E, Esposito L, Mistrangelo M, Rebecchi F, Arezzo A, Morino M. Analysis of Early and Long-Term Oncologic Outcomes After Converted Laparoscopic Resection Compared to Primary Open Surgery for Rectal Cancer. World J Surg. 2018 Oct;42(10):3405-3414. doi: 10.1007/s00268-018-4614-x. PMID 29610930
- [Background] de Neree Tot Babberich MPM, van Groningen JT, Dekker E, Wiggers T, Wouters MWJM, Bemelman WA, Tanis PJ; Dutch Surgical Colorectal Audit. Laparoscopic conversion in colorectal cancer surgery; is there any improvement over time at a population level? Surg Endosc. 2018 Jul;32(7):3234-3246. doi: 10.1007/s00464-018-6042-2. Epub 2018 Jan 17. PMID 29344789
- See also: Society of American Gastrointestinal and and Endoscopic Surgeons, Guidelines for Laparoscopic resection of curable colon and rectal cancer, Guidelines. (2015) — http://www.sages.org/publications/guidelines/guidelines